CLINICAL TRIAL: NCT00098059
Title: A Multicenter, Open-label, Single-arm, Two-step Study to Evaluate the Safety and Single-dose Pharmacokinetics of Famciclovir and Multiple-dose Safety After Administration of Famciclovir Oral Pediatric Formulation to Children 1 to 12 Years of Age With Herpes Simplex Infection
Brief Title: Famciclovir Pediatric Formulation in Children 1 to 12 Years of Age With Herpes Simplex Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFAM810B2303
Record Dates: First submitted 2004-12-02; First posted 2004-12-03 (Estimated); Results first posted 2009-05-06 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Herpes Simplex
Keywords: herpes simplex; cold sores; fever blisters; children; Famvir; famciclovir
MeSH Terms: conditions — Herpes Simplex; Herpes Labialis | interventions — Famciclovir

ARMS (1):
- Famciclovir, pediatric oral formulation (Experimental): single-arm
  Interventions: Drug: Famciclovir

INTERVENTIONS:
Drug: Famciclovir — Famciclovir sprinkle capsules, 25 mg and 100 mg, using OraSweet® syrup vehicle

SUMMARY:
This study will evaluate the safety and blood levels of a new pediatric formulation of Famvir in children 1-12 years of age. In Part A, patients will receive a single dose of famciclovir (12.5 mg/kg) to assess pharmacokinetics (PK) and safety. In Part B, patients will receive multiple doses of famciclovir alone or with concomitant oral anti-herpes therapy to assess safety and tolerability. Part B will start only after PK data from Part A had been analyzed.

ELIGIBILITY:
Inclusion Criteria:

* History or laboratory evidence of herpes simplex infection
* Clinical evidence or suspicion of herpes simplex infection

Exclusion Criteria:

* Patients unable to swallow
* Concomitant use of probenecid
* Positive pregnancy test

Additional protocol-defined inclusion/exclusion criteria may apply. For detailed information on eligibility, please contact the study center nearest to you or call the following numbers: 1-862-778-3544 or 1-434-951-3228

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2005-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Children's Hospital, Denver, Colorado
  - Children's Memorial Hospital, Chicago, Illinois
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Columbia University Medical Center, New York, New York
  - State University of New York at, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Children's Medical Center of Dallas, Dallas, Texas
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
- Panama (2):
  - Panama Minister of Health, David, Chiriquí Province
  - Panama Minister of Health, Panama City

REFERENCES:
- [Derived] Saez-Llorens X, Yogev R, Arguedas A, Rodriguez A, Spigarelli MG, De Leon Castrejon T, Bomgaars L, Roberts M, Abrams B, Zhou W, Looby M, Kaiser G, Hamed K. Pharmacokinetics and safety of famciclovir in children with herpes simplex or varicella-zoster virus infection. Antimicrob Agents Chemother. 2009 May;53(5):1912-20. doi: 10.1128/AAC.01054-08. Epub 2009 Mar 9. PMID 19273678

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A (Single-dose of Famciclovir): Includes 27 patients enrolled in Part A. Two adolescent patients (13 to 18 years) were enrolled in Part A of this study under an amendment to the protocol to include adolescent aged patients. The amendment was rescinded in compliance with an FDA Pediatric Written Request and no further adolescent aged patients were enrolled.
- Part B (Multiple-dose of Famciclovir): Includes 47 patients enrolled in Part B. Part B started only after pharmacokinetic (PK) data from Part A had been analyzed. One patient that participated in Part A of the study also participated in Part B.
Period: Overall Study
Arm/Group | Part A (Single-dose of Famciclovir) | Part B (Multiple-dose of Famciclovir)
Started | 27 | 47
Completed | 27 | 46
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part A (Single-dose of Famciclovir): Each patient in Part A received a single dose of famciclovir (12.5 mg/kg).
- Part B (Multiple-dose of Famciclovir): Each patient in Part B received famciclovir twice a day (b.i.d.) approximately 12 hours apart for 7 days for a total of 14 doses. An 8-step dosing scheme (ranged from 150 mg b.i.d. to 500 mg b.i.d.) was used to determine the weight-based adjusted daily dose.
- Total: Total of all reporting groups
Arm/Group | Part A (Single-dose of Famciclovir) | Part B (Multiple-dose of Famciclovir) | Total
Number analyzed (Participants) | 27 | 47 | 74
Age, Customized [Number; unit: participants]
  1 to <2 years | 4 | 13 | 17
  2 to <6 years | 13 | 16 | 29
  6 to <=12 years | 8 | 18 | 26
  13 to <=18 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 41
  Male | 10 | 23 | 33

OUTCOME MEASURES:

1. Secondary Outcome: Overall Acceptability of Pediatric Oral Formulation by Patients in Part A of the Study.
Description: Overall acceptability of the study medication was determined by caretaker response.
Time Frame: Day 1, after swallowing the dose.
Population: Includes all 27 patients enrolled in Part A of the study.
Measure: Number; unit: participants
Arm/Group | 1 to < 2 Years | 2 to <6 Years | 6 to <13 Years | 13 to <=18 Years
Number analyzed (Participants) | 4 | 13 | 8 | 2
participants
  Badly | 1 | 4 | 0 | 2
  Neither bad nor good | 1 | 1 | 4 | 0
  Well | 2 | 8 | 4 | 0

2. Secondary Outcome: Overall Acceptability of Pediatric Oral Formulation by Patients in Part B of the Study.
Description: Overall acceptability of the study medication was determined by caretaker response.
Time Frame: Day 1 at clinic: after swallowing first dose
Population: Includes all 47 patients enrolled in Part B of the study.
Measure: Number; unit: participants
Arm/Group | 1 to < 2 Years | 2 to <6 Years | 6 to <13 Years | 13 to <=18 Years
Number analyzed (Participants) | 13 | 16 | 18 | 0
participants
  Badly | 9 | 6 | 7 |
  Neither bad nor good | 2 | 1 | 2 |
  Well | 2 | 9 | 9 |

3. Secondary Outcome: Overall Acceptability of Pediatric Oral Formulation by Patients in Part B of the Study
Description: Overall acceptability of study medication was determined by caretaker response.
Time Frame: Day 8 at home: after swallowing last dose
Population: Includes all 47 patients enrolled in Part B of the study. Response was not available for 1 patient in the 2 to <6 years and 6 to <=12 years groups.
Measure: Number; unit: participants
Arm/Group | 1 to < 2 Years | 2 to <6 Years | 6 to <13 Years | 13 to <=18 Years
Number analyzed (Participants) | 13 | 16 | 18 | 0
participants
  Badly | 7 | 5 | 3 |
  Neither bad nor good | 3 | 3 | 3 |
  Well | 3 | 7 | 11 |

4. Primary Outcome: Safety and Tolerability of a Single-dose of Famciclovir in Part A of the Study.
Description: A patient with multiple adverse events (AEs) within the primary system organ class is counted only once in total row.
Time Frame: 8 hours and 24 hours after study drug administration (Part A)
Population: Includes all 27 patients enrolled in Part A of the study.
Measure: Number; unit: participants
Arm/Group | 1 to < 2 Years | 2 to <6 Years | 6 to <=12 Years | 13 to <= 18 Years
Number analyzed (Participants) | 4 | 13 | 8 | 2
participants
  Patients with AEs | 0 | 2 | 1 | 2
  Gastrointestinal disorders | 0 | 1 | 0 | 1
  Nervous system disorders | 0 | 0 | 1 | 1
  General disorders and administration site | 0 | 0 | 0 | 1
  Infections and infestations | 0 | 1 | 0 | 0
  Skin and subcutaneous tissue disorders | 0 | 1 | 0 | 0

5. Primary Outcome: Maximum Observed Plasma Concentration of Penciclovir (Cmax)
Description: PK parameter; penciclovir is the active metabolite of famciclovir.
Time Frame: plasma level measurements: pre-dose, 1, 2, 3, 4 and 5 hours post-dose
Population: Includes all 27 patients enrolled in Part A of the study.
Measure: Mean (Full Range); unit: μg/mL
Arm/Group | 1 to < 2 Years | 2 to <6 Years | 6 to <=12 Years | 13 to <= 18 Years
Number analyzed (Participants) | 4 | 13 | 8 | 2
μg/mL | 2.84 (1.25) [1.42 to 4.47] | 2.44 (0.94) [0.42 to 3.81] | 2.82 (0.65) [1.52 to 3.79] | 1.89 [1.06 to 2.72]

6. Primary Outcome: Time of Maximum Observed Plasma Concentration of Penciclovir (Tmax)
Description: PK parameter; penciclovir is the active metabolite of famciclovir.
Time Frame: Plasma level measurements: pre-dose, 1, 2, 3, 4 and 5 hours post-dose
Population: Includes all 27 patients enrolled in Part A of the study.
Measure: Median (Full Range); unit: hours
Arm/Group | 1 to < 2 Years | 2 to <6 Years | 6 to <=12 Years | 13 to < =18 Years
Number analyzed (Participants) | 4 | 13 | 8 | 2
hours | 1.21 [1.00 to 1.50] | 1.07 [1.00 to 4.03] | 1.00 [1.00 to 2.07] | 1.47 [0.97 to 1.97]

7. Primary Outcome: Area Under the Penciclovir Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-∞)
Description: PK parameter; penciclovir is the active metabolite of famciclovir.
Time Frame: Plasma level measurements: pre-dose, 1, 2, 3, 4 and 5 hours post-dose
Population: Includes 26 of 27 patients enrolled in Part A of the study.
Measure: Mean (Full Range); unit: (μg/mL)h
Arm/Group | 1 to < 2 Years | 2 to <6 Years | 6 to <=12 Years | 13 to <= 18 Years
Number analyzed (Participants) | 4 | 12 | 8 | 2
(μg/mL)h | 6.17 (2.42) [3.43 to 8.99] | 6.85 (1.55) [3.19 to 9.12] | 8.15 (1.01) [6.49 to 9.71] | 5.93 (0) [4.84 to 7.01]

8. Primary Outcome: Apparent Oral Clearance of Penciclovir (CL/F)
Description: PK parameter; penciclovir is the active metabolite of famciclovir.
Time Frame: Plasma level measurements: pre-dose, 1, 2, 3, 4 and 5 hours post-dose
Population: Includes 26 of 27 patients enrolled in Part A of the study.
Measure: Mean (Full Range); unit: L/h
Arm/Group | 1 to < 2 Years | 2 to <6 Years | 6 to <=12 Years | 13 to <= 18 Years
Number analyzed (Participants) | 4 | 12 | 8 | 2
L/h | 20.8 (8.5) [11.0 to 28.8] | 25.1 (4.3) [18.1 to 33.3] | 43.7 (9.6) [32.4 to 60.8] | 68.8 (0) [56.2 to 81.5]

9. Primary Outcome: Apparent Terminal Elimination Half-life of Penciclovir (T1/2)
Description: PK parameter; penciclovir is the active metabolite of famciclovir
Time Frame: Plasma level measurements: pre-dose, 1, 2, 3, 4 and 5 hours post-dose
Population: Includes 26 of 27 patients enrolled in Part A of the study.
Measure: Mean (Full Range); unit: hours
Arm/Group | 1 to < 2 Years | 2 to <6 Years | 6 to <=12 Years | 13 to <= 18 Years
Number analyzed (Participants) | 4 | 12 | 8 | 2
hours | 1.09 (0.08) [1.01 to 1.18] | 1.36 (0.20) [1.10 to 1.70] | 1.60 (0.25) [1.30 to 2.11] | 1.86 [1.60 to 2.12]

10. Primary Outcome: Safety and Tolerability of Famciclovir Pediatric Oral Formulation in Part B of the Study.
Description: A patient with multiple AEs within the primary system organ class is counted only once in total row.
Time Frame: Administered 2 times daily over 7 days
Population: Includes 47 patients enrolled in Part B of the study.
Measure: Number; unit: participants
Arm/Group | 1 to < 2 Years | 2 to <6 Years | 6 to <13 Years | 13 to <=18 Years
Number analyzed (Participants) | 13 | 16 | 18 | 0
participants
  Patients with AEs | 6 | 8 | 12 |
  Gastrointestinal disorders | 4 | 3 | 6 |
  Nervous system disorders | 0 | 2 | 5 |
  General disorders and administration site | 3 | 1 | 1 |
  Respiratory, thoracic and mediastinal disorders | 1 | 1 | 2 |
  Infections and infestations | 3 | 0 | 0 |
  Skin and subcutaneous tissue disorders | 1 | 2 | 0 |
  Vascular disorders | 0 | 0 | 2 |
  Injury, poisoning and procedural complications | 0 | 1 | 1 |
  Investigations | 1 | 0 | 0 |
  Metabolism and nutrition disorders | 1 | 0 | 0 |

ADVERSE EVENTS:
Time Frame: Patients in Parts A and B of the study who experienced adverse events. These AEs are presented by system organ class for each age group in the safety population.
Arm/Group | Part A (Single-dose of Famciclovir) | Part B (Multiple-dose of Famciclovir)
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/47
Other Adverse Events (participants affected / at risk) | 5/27 | 23/47
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (Single-dose of Famciclovir) (N=27) | Part B (Multiple-dose of Famciclovir) (N=47)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 4
Pyrexia (General disorders) | 1 | 2
Furuncle (Infections and infestations) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 5
Diarrhea (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.